CLINICAL TRIAL: NCT07062159
Title: Effectiveness of Psychoeducational Intervention in Reducing Postpartum Depressive Symptoms and Strengthening Mother-Infant Bonding: A Randomized Controlled Trial From the Watson Model Perspective
Brief Title: Psychoeducational Intervention to Reduce Depressive Symptoms and Strengthen Mother-Infant Bonding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yasemin Ozhuner (Other)
Responsible Party: Sponsor-Investigator, Yasemin Ozhuner, DR, Eskisehir Osmangazi University
Organization: Eskisehir Osmangazi University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Attachment and depression
Record Dates: First submitted 2025-07-02; First posted 2025-07-14 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Postpartum Depression; Psychoeducation; Mother-Infant Interaction
Keywords: Postpartum Depression; Watson model; psychoeducation; Mother-Infant Interaction
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: The pregnant women included in the sample were informed about the study and their written consent was obtained. Six interviews were conducted with the pregnant women, four at one-week intervals before birth and one on the seventh day and fourth week after birth. These interviews were conducted with the women one-on-one and face-to-face. The women in the control group did not receive any treatment other than routine care at family health centers. The psychoeducation program was administered to the women in the intervention group in six interviews.
Masking Description: control group (44)
  intervention group (44)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Active Comparator): Active Comparator: intervention group The pregnant women in the sample were informed about the study and their written consent was obtained. A total of six interviews were conducted with the pregnant women, four at one-week intervals before birth and one interview on the seventh day and fourth week after birth. These interviews were conducted with the women one-on-one and face-to-face. The psychoeducation program was applied to the women in the intervention group in six interviews. In the first interview, the women were given a booklet of the psychoeducation intervention program based on the Watson Human Caring Model for postpartum care and the interview was conducted within the scope of the program. The psychoeducation intervention program interviews based on the Watson Human Caring Model in the study were conducted according to the Watson Human Caring Model improvement processes and psychoeducation techniques. The interviews lasted between 60-90 minutes on average.
  Interventions: Other: the psychoeducation intervention program
- control group (Placebo Comparator): Placebo Comparator: Control Group The pregnant women in the sample were informed about the study and their written consent was obtained. Six interviews were conducted with the pregnant women, four at one-week intervals before delivery and once on the seventh day and fourth week after delivery. These interviews were conducted with the women one-on-one and face-to-face. The women in the control group did not receive any treatment other than their routine care at family health centers. In routine care, pregnant women were examined for edema, varicose veins, weight, blood pressure, pulse, laboratory findings, baby heart sounds, medication intake, chronic disease follow-up and vaccination. Pregnant women were provided with counseling if they had any questions. After delivery, women were provided with medication intake, blood pressure, fever, pulse, bleeding and laboratory findings and counseling if they had any questions.
  Interventions: Other: routine care

INTERVENTIONS:
Other: the psychoeducation intervention program — The content of the psychoeducation intervention program based on the Watson Human Caring Model will consist of the postpartum process and care, maternal blues, postpartum psychosis, postpartum depression, frequency, causes, predisposing factors, symptoms, effects on mother, child and community health, diagnosis and treatment, preventive practices, social support, adaptation to the role of motherhood, mother and baby bonding, practices that will strengthen mother-baby bonding, breast milk and breastfeeding, nutrition and baby care, problems encountered in baby care and solution suggestions.
  Arms: intervention group
Other: routine care — routine care
  Arms: control group

SUMMARY:
The study aims to evaluate the effectiveness of a psychoeducational intervention designed within the framework of the Watson Human Caring Model in reducing postpartum depressive symptoms and creating a stronger mother-infant bond. Specifically, it aims to investigate whether a person-centered approach based on the principles of Watson's caring science can significantly increase the psychological well-being of postpartum mothers and improve the quality of their relationship with their babies.

DETAILED DESCRIPTION:
The pregnant women included in the sample were informed about the study and their written consent was obtained. Six interviews were conducted with the pregnant women, four at one-week intervals before birth and one on the seventh day and fourth week after birth. These interviews were conducted with the women one-on-one and face-to-face. The women in the control group did not receive any treatment other than routine care at family health centers. The psychoeducation program was applied to the women in the intervention group in six interviews.

ELIGIBILITY:
Inclusion Criteria:

* • Women in their 20-35th week of pregnancy,

  * Volunteers,
  * Over 18 years of age,
  * Literate,
  * No visual, hearing or mental disabilities,
  * Having a healthy baby weighing over 2500 grams,
  * Being in the same environment with their baby after birth,
  * Having a healthy fetus on ultrasound will be included in the study.

Exclusion Criteria:

* • Those diagnosed with depression or other mental illnesses by a physician,

  * Those taking medication for mental illness,
  * Women who have given birth prematurely,
  * Stillbirth,
  * Those who have not participated in more than one interview will not be included in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2025-07-02 (Actual); Primary Completion 2025-08-19 (Actual); Study Completion 2026-01-05 (Actual)

PRIMARY OUTCOMES:
Prenatal Attachment Scale | 1 day (first meeting during pregnancy)
  Prenatal Attachment Scale The scale consists of 21 items in total. The highest score on the scale is 84, the lowest score is 21, and the increase in the total score obtained from the scale indicates that prenatal attachment is positive.
Edinburgh Postpartum Depression Scale | 1 day (first meeting during pregnancy and at the fourth week postpartum)
  It is a 10-item self-report scale that measures maternal depressive symptoms over the past seven days. Higher scores reflect more depressive symptoms. Symptoms are rated on a 4-point Likert scale with scores ranging from 0 to 30. The cut-off score of the scale was determined as ≥13. If the total score of the scale is 12 or less, the participant is not at risk for PPD, but if he scores 13 or more, he is at risk.
Mother-Infant Attachment Scale | fourth week postpartum
  Mother-Infant Attachment Scale This scale, which is used from the first day after birth, allows the mother to describe her feelings towards her baby in one word. The lowest score that can be obtained from the scale is 0 and the highest score is 24. As the score increases, attachment is negatively affected.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Özhüner, Principal Investigator — Eskişehir Vadişehir Family center odunpazarı Turkey; Nebahat Ozerdogan, Study Director — Eskisehir Osmangazi University odunpazarı turkey
Locations (1):
- Eskisehir Osmangazi University, Eskişehir, Odunpazarı, Turkey (Türkiye)